CLINICAL TRIAL: NCT00022763
Title: A Phase I/II Pharmacokinetic and Safety Study of T-20 in Combination With an Optimized Background in HIV Infected Children and Adolescents
Brief Title: T-20 Plus a Selected Anti-HIV Treatment in HIV-Infected Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV16056; T20-310; 295E
Record Dates: First submitted 2001-08-11; First posted 2001-08-31 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: HIV Infections
Keywords: Anti-HIV Agents; pentafuside
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide

SUMMARY:
This study will evaluate T-20 in children.

DETAILED DESCRIPTION:
Children are stratified by age group (3 through 11 years and 12 through 16 years). Samples for HIV-1 genotype and phenotype resistance testing are obtained at screening to aid in the selection of concomitant antiretrovirals. Simultaneous to initiating T-20, all patients begin a "new" optimized antiretroviral regimen based on the patients' prior treatment history, historical resistance testing results, and the results of the testing performed at screening. Patients are followed for safety and other assessments at Weeks 1, 2, and 4, then monthly through Week 24 and bimonthly through Week 48. Pharmacokinetic sampling at selected study visits are performed.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 3 through 16 years of age and have the consent of parent or guardian.
* Have a viral load of at least 5000 copies/ml.
* Have taken at least 2 of the 3 licensed anti-HIV drug classes for at least 3 months.
* Have been on stable therapy for at least 4 weeks.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2001-08; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Children's Hosp Los Angeles, Los Angeles, California
  - Univ of Florida Gainesville, Gainesville, Florida
  - New York Hosp - Cornell / Program for Children with AIDS, New York, New York
  - Mount Sinai Hosp, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Children's Hosp of the King's Daughters, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 52 participants were enrolled in this study conducted at 16 centers in Spain and United States between 23 August 2001 and 09 December 2004.
Groups:
- Stratum A: Participants of age greater than or equal to (>=) 3 years and less than 12 years received enfuvirtide subcutaneously twice daily (BID) at 2.0 mg/kg per dose, up to the adult maximum of 90 mg per dose for 48 weeks. At the end of the 48 weeks of treatment, participants were allowed to continue into the extension phase and take enfuvirtide up to a maximum of an additional 48 weeks (a total of 96 weeks from study entry), or until 12 weeks after the commercial availability of enfuvirtide in the country of the participant's participation, whichever came first.
- Stratum B: Participants of age >= 12 years and less than 17 years received enfuvirtide subcutaneously BID at 2.0 mg/kg per dose, up to the adult maximum of 90 mg per dose for 48 weeks. At the end of the 48 weeks of treatment, participants were allowed to continue into the extension phase and take enfuvirtide up to a maximum of an additional 48 weeks (a total of 96 weeks from study entry), or until 12 weeks after the commercial availability of enfuvirtide in the country of the participant's participation, whichever came first.
Period: Overall Study
Arm/Group | Stratum A | Stratum B
Started | 24 | 28
Completed | 15 | 11
Not Completed | 9 | 17
Not completed — Adverse Event | 1 | 2
Not completed — Injection Site Reactions | 0 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Insufficient Therapy | 1 | 0
Not completed — Admin | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Stratum A: Participants of age >= 3 years and less than 12 years received enfuvirtide subcutaneously BID at 2.0 mg/kg per dose, up to the adult maximum of 90 mg per dose for 48 weeks. At the end of the 48 weeks of treatment, participants were allowed to continue into the extension phase and take enfuvirtide up to a maximum of an additional 48 weeks (a total of 96 weeks from study entry), or until 12 weeks after the commercial availability of enfuvirtide in the country of the participant's participation, whichever came first.
- Total: Total of all reporting groups
Arm/Group | Stratum A | Stratum B | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (1.8) | 13.9 (1.6) | 11.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 9 | 19 | 28

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) From 0-12 Hours for Enfuvirtide and Its Metabolite (Ro 50-6343)
Description: The Area Under the Plasma Concentration-Time Curve (AUC) is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption. AUC was calculated from plasma concentration-time data (on Day 7) using standard non-compartmental pharmacokinetic methods.
Time Frame: Pre-dose (time 0), and 2, 4, 8, and 12 hours post-dose (Week 1)
Population: Intensive PK Analysis Population: The first 12 participants enrolled per age group and all children aged 3 to 6 years who underwent intensive pharmacokinetic sampling at week 1 were included within the intensive PK analysis population.
Measure: Mean (Standard Deviation); unit: microgram hour per milliliter (mcg.h/mL)
Groups:
- Stratum A: Participants of age >= 3 years and less than 12 years received enfuvirtide subcutaneously twice daily (BID) at 2.0 mg/kg per dose, up to the adult maximum of 90 mg per dose for 48 weeks. At the end of the 48 weeks of treatment, participants were allowed to continue into the extension phase and take enfuvirtide up to a maximum of an additional 48 weeks (a total of 96 weeks from study entry), or until 12 weeks after the commercial availability of enfuvirtide in the country of the participant's participation, whichever came first.
- Stratum B: Participants of age >= 12 years and less than 17 years received enfuvirtide subcutaneously twice daily (BID) at 2.0 mg/kg per dose, up to the adult maximum of 90 mg per dose for 48 weeks. At the end of the 48 weeks of treatment, participants were allowed to continue into the extension phase and take enfuvirtide up to a maximum of an additional 48 weeks (a total of 96 weeks from study entry), or until 12 weeks after the commercial availability of enfuvirtide in the country of the participant's participation, whichever came first.
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 12 | 13
microgram hour per milliliter (mcg.h/mL)
  Enfuvirtide | 56.1 (19.4) | 52.7 (27.4)
  Metabolite (Ro 50-6343) | 3.07 (2.77) | 3.41 (2.09)

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Enfuvirtide and Its Metabolite (Ro 50-6343)
Description: The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration. Cmax was calculated from plasma concentration-time data (on Day 7) using standard non-compartmental pharmacokinetic methods.
Time Frame: Pre-dose (time 0), and 2, 4, 8, and 12 hours post-dose (Week 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 12 | 13
mcg/mL
  Enfuvirtide | 6.43 (2.15) | 5.88 (2.81)
  Metabolite (Ro 50-6343) | 0.434 (0.667) | 0.450 (0.341)

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Enfuvirtide
Description: Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time Frame: Pre-dose (time 0), and 2, 4, 8, and 12 hours post-dose (Week 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 12 | 13
hour | 4.13 (1.35) | 5.05 (2.67)

4. Secondary Outcome: Minimum Plasma Concentration (Ctrough) for Enfuvirtide and Its Metabolite (Ro 50-6343)
Description: Ctrough is defined as the lowest concentration that a drug reaches before the next dose is administered.
Time Frame: Pre-dose (time 0), and 2, 4, 8, and 12 hours post-dose (Week 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 12 | 13
mcg/mL
  Enfuvirtide | 2.87 (1.49) | 2.98 (1.66)
  Metabolite (Ro 50-6343) | 0.177 (0.089) | 0.242 (0.146)

5. Secondary Outcome: AUC12h Ratio of Enfuvirtide Metabolite (Ro 50-6343)/ENF (Ro 29-9800)
Description: The ratio of the area under plasma concentration-time curve from time 0 to 12 hours of Enfuvirtide Metabolite (Ro 50-6343) versus enfuvirtide was calculated.
Time Frame: Pre-dose (time 0), and 2, 4, 8, and 12 hours post-dose (Week 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 12 | 13
Ratio | 5.31 (3.55) | 7.12 (3.98)

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event.
Time Frame: Up to Week 4 after discontinuation of therapy
Population: Safety Analysis Population: All participants who received at least one dose of study medication were included.
Measure: Number; unit: participants
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 24 | 28
participants
  Any AE | 24 | 25
  Any SAE | 8 | 15

7. Secondary Outcome: Number of Participants With Treatment Emergent Grade 3 or Grade 4 Laboratory Abnormalities
Description: Pediatric AIDS Clinical Trials Group (PACTG) toxicity grading scale was used for reviewing and grading clinically significant laboratory abnormalities. PACTG Grade 3 and Grade 4 were considered Severe and life threatening, respectively.
Time Frame: Up to Week 96
Population: Safety Analysis Population: All participants who received at least one dose of study medication were included.
Measure: Number; unit: participants
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 24 | 26
participants
  Platelets Grade 3 | 0 | 2
  Platelets Grade 4 | 1 | 0
  Neutrophils Grade 3 | 0 | 0
  Neutrophils Grade 4 | 1 | 0
  ASAT Grade 3 | 2 | 0
  ASAT Grade 4 | 0 | 0
  ALAT Grade 3 | 1 | 0
  ALAT Grade 4 | 0 | 0
  Total Bilirubin Grade 3 | 0 | 1
  Total Bilirubin Grade 4 | 0 | 0
  GGT Grade 3 | 0 | 1
  GGT Grade 4 | 0 | 0
  Amylase Grade 3 | 1 | 1
  Amylase Grade 4 | 1 | 1

8. Secondary Outcome: Number of Participants Who Died
Time Frame: Up to Week 96
Population: Safety Analysis Population: All participants who received at least one dose of study medication were included.
Measure: Number; unit: participants
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 24 | 28
participants | 1 | 1

9. Secondary Outcome: Number of Participants Who Prematurely Withdrew Due to AE
Time Frame: Up to Week 96
Population: Safety Analysis Population: All participants who received at least one dose of study medication were included.
Measure: Number; unit: participants
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 24 | 28
participants | 9 | 17

10. Secondary Outcome: Number of Participants With Worst Local Injection Site Reactions
Description: Numbers of Participants With worst local injection site reactions were reported. Localized injection site reactions like erythema, induration, pruritus, nodule and cyst, and ecchymosis were recorded.
Time Frame: Up to Week 96
Population: Safety Analysis Population: All participants who received at least one dose of study medication were included.
Measure: Number; unit: participants
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 24 | 28
participants
  Erythema | 13 | 19
  Nodules and Cysts | 16 | 14
  Induration | 21 | 20
  Pruritus | 10 | 9
  Ecchymosis | 6 | 8
  Others | 5 | 10

ADVERSE EVENTS:
Time Frame: Up to Week 96
Description: All participants who received at least one dose of study medication were included in safety analysis.
Groups:
- Enfuvirtide: Participants in stratum A (age >= 3 years and less than 12 years received Enfuvirtide Subcutaneously BID at 2.0 mg/kg per dose, up to the adult maximum of 90 mg per dose) and in stratum B (age >= 12 years and less than 17 years received Enfuvirtide Subcutaneously BID at 2.0 mg/kg per dose, up to the adult maximum of 90 mg per dose).
Arm/Group | Enfuvirtide
Serious Adverse Events (participants affected / at risk) | 31/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enfuvirtide (N=52)
Pneumonia nos (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 3
Gastroenteritis nos (Infections and infestations) | 2
Bronchiolitis (Infections and infestations) | 1
Bronchitis nos (Infections and infestations) | 1
Colitis pseudomembranous (Infections and infestations) | 1
Gastroenteritis viral nos (Infections and infestations) | 1
Kawasaki's disease (Infections and infestations) | 1
Lobar pneumonia nos (Infections and infestations) | 1
Pneumonia viral nos (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis nos (Infections and infestations) | 1
Staphylococcal abscess (Infections and infestations) | 1
Pyrexia (General disorders) | 2
Injection site abscess (General disorders) | 1
Multi-organ failure (General disorders) | 1
Metabolic disorder nos (Metabolism and nutrition disorders) | 1
Tetany (Metabolism and nutrition disorders) | 1
Blood creatinine increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dystonia (Nervous system disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enfuvirtide (N=52)
Upper respiratory tract infection nos (Infections and infestations) | 22
Otitis media nos (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 9
Sinusitis nos (Infections and infestations) | 8
Oral candidiasis (Infections and infestations) | 6
Body tinea (Infections and infestations) | 4
Impetigo nos (Infections and infestations) | 4
Viral infection nos (Infections and infestations) | 4
Gastroenteritis nos (Infections and infestations) | 3
Herpes simplex (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Bronchospasm nos (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Rhinitis allergic nos (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Asthma nos (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Vomiting nos (Gastrointestinal disorders) | 11
Diarrhoea nos (Gastrointestinal disorders) | 9
Abdominal pain nos (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Loose stools (Gastrointestinal disorders) | 5
Sore throat nos (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 3
Dermatitis Nos (Skin and subcutaneous tissue disorders) | 10
Acne Nos (Skin and subcutaneous tissue disorders) | 5
Eczema Seborrhoeic (Skin and subcutaneous tissue disorders) | 3
Rash papular (Skin and subcutaneous tissue disorders) | 3
Pyrexia (General disorders) | 11
Fatigue (General disorders) | 6
Conjunctivitis nec (Eye disorders) | 5
Conjunctivitis allergic (Eye disorders) | 4
Vision blurred (Eye disorders) | 3
Weight decreased (Investigations) | 5
Haematuria present (Investigations) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Headache Nos (Nervous system disorders) | 6
Hypersensitivity Nos (Immune system disorders) | 4
Earache (Ear and labyrinth disorders) | 3
Arthropod bite (Injury, poisoning and procedural complications) | 3
Appetite decreased nos (Metabolism and nutrition disorders) | 3
Dysuria (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.